CLINICAL TRIAL: NCT01250002
Title: The Effect of Perioperative Systemic Lidocaine on Quality of Recovery After Outpatient Gynecologic Laparoscopy
Brief Title: Lidocaine and Outpatient Gynecologic Laparoscopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Gildasio De Oliveira, Gildasio De Oliveira, M.D. Principal Investigator, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: STU00025240
Record Dates: First submitted 2010-11-27; First posted 2010-11-30 (Estimated); Results first posted 2013-06-21 (Estimated); Last update posted 2014-06-26 (Estimated); Status verified 2014-06

CONDITIONS: Pain
Keywords: Pain; MQOR 40; Lidocaine; Gynecologic; Surgery; Laparoscopic
MeSH Terms: conditions — Pain | interventions — Lidocaine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lidocaine (Active Comparator): Lidocaine administration 1.5 mg/kg bolus followed by a 2 mg/kg/hr infusion via intravenous catheter
  Interventions: Drug: Lidocaine
- Placebo (Placebo Comparator): Placebo will receive the same volume of saline infusion.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Placebo — Placebo will receive the same volume of saline infusion.
  Arms: Placebo
Drug: Lidocaine — Lidocaine administration 1.5 mg/kg bolus followed by a 2 mg/kg/hr infusion via intravenous catheter
  Arms: Lidocaine

SUMMARY:
Although ambulatory gynecological laparoscopy is considered to be a minimally invasive surgical procedure, only 60% of patients undergoing this procedure are satisfied with postoperative pain control. Postoperative pain can lead to physiological, immunological and psychological derangements in patients.It also has been shown to be the most common cause of hospital admission after outpatient surgery.

Opioids constitute the most commonly used pain management strategy after surgery, however they have many undesirable side effects including nausea, vomiting and respiratory depression. Different strategies have been developed to decrease the amount of opioid required after surgery. Opioid sparing drugs as well as regional anesthesia have been shown to be effective. Systemic administration of lidocaine has been shown to decrease opioid consumption, improve recovery of bowel function and promote a better recovery after inpatient procedures. Lidocaine has been shown to have analgesic, antihyperalgesic and anti-inflammatory properties. It also has an excellent safety profile when give by a low-dose infusion.

The improvement of surgical technique and anesthesia care has made major adverse outcomes infrequent, especially in the ambulatory setting. Assessing patient's quality of recovery has become an important outcome in several studies. The patient's capacity to return to his normal activities is one of the most important sign of a successful outpatient procedure and it has significant economic implications.

Quality of recovery -40(QoR-40) is a validated 40 item instrument to assess the quality of post-operative recovery. Myels et al. have concluded that the QoR-40 would be a useful outcome measure to assess the impact on changes in health care delivery, but anesthesia studies underutilize this instrument.

The research question for the study is; does the use of systemic perioperative lidocaine improve quality of recovery after outpatient laparoscopy?

DETAILED DESCRIPTION:
70 subjects will be randomly allocated into 2 groups, using a computer generated table of random numbers. Group A (study group) will receive lidocaine. Group B (control group) will receive the same volume of saline infusion. The study drugs will be prepared by one of the investigators in the study. Subjects will be recruited up to 21 days prior to surgery.They will be premedicated with intravenous (IV) midazolam 0.04 mg/kg. Routine ASA monitors will be applied. Anesthesia will be induced with remifentanil infusion started at 0.1 mcg/kg/minute titrated to keep blood pressure within 20% of the baseline and propofol 1.0 -2.0 mg/kg. Group A will receive lidocaine 1.5mg/kg bolus and Group B the equivalent volume of saline. Subjects will be monitored with a 5 lead EKG throughout the lidocaine administration and if any arrhythmia is detected. The study drug will be stopped and investigators unblinded.

Tracheal intubation will be facilitated with rocuronium (0.6 mg/kg) or succinylcholine (1-2mg /kg). Immediately after the induction, group A will receive lidocaine infusion (2 mg/kg/hr IV). Group B will receive the equivalent volume of saline; both infusions will be continued until 1 hour after arrival in the PACU. Anesthesia will be maintained with desflurane titrated to maintain a bispectral index (BIS) between 40-60 , remifentanil infusion started at 0.1mcg/kg/min titrated to keep blood pressure within 20 % of baseline values , and rocuronium that will be administered at the discretion of the anesthesiologist. Upon termination of the surgery, neuromuscular blockade will be antagonized with a combination of neostigmine 0.05mg/kg and glycopyrrolate 0.01 mg/kg. Ondansetron 4 mg IV will be administered to prevent postoperative nausea and vomiting. Subject will be evaluated for pain in the OR after extubation, using a numeric rating scale, if pain greater than 4/10 they will receive hydromorphone (10 mcg/kg IV). In PACU, subjects will receive IV hydromorphone in divided doses as needed to achieve a verbal rating score for pain <4 out of 10 and they will be evaluated every 15 minutes .They will also receive metoclopramide (20 mg IV ) as rescue antiemetic in PACU. Discharge readiness will be assessed by a PACU nurse using the modified Post Anesthesia Discharge Scoring System (MPADSS) score every 15 minutes for about 3 hours or until ready for discharge.The primary and secondary outcomes will be assessed by an independent observer who will be blinded to group allocation. Study personnel will contact the subject at 24 hours to assess well being, (nausea, vomiting and opioid consumption. Subject will be contacted by telephone by the study staff and will complete the Modified Quality of Recovery 40 (MQOR40) at 24 hours post surgery.

ELIGIBILITY:
Inclusion Criteria:

* Female patients undergoing outpatient laparoscopic gynecologic surgery
* American society of anesthesiologists class (ASA) Physical status (PS) I and II
* Age between 18 and 64 years
* Fluent in English
* Body mass index (BMI) less than 35

Exclusion Criteria:

* History of allergy to local anesthetics
* History of chronic opioid use
* Pregnant patients
* Body Mass Index (BMI) greater than 35
* History of electrocardiogram (EKG) abnormalities
* Hepatic Impairment
* History of congestive heart failure
* Electrocardiogram (EKG) abnormalities
* History of heart block (subject with history of heart block)
* Current use of anti-arrhythmic medications

Drop -Outs:

* Patient or surgeon request
* Conversion of the surgery from laparoscopic to open

Ages: 18 Years to 64 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 70 (Actual)
Dates: Start 2010-11; Primary Completion 2011-09 (Actual); Study Completion 2011-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gildasio De Oliveira, MD, Principal Investigator — Northwestern University
Locations (1):
- Prentice Womens Hospital, Chicago, Illinois, United States

REFERENCES:
- [Background] Lovatsis D, Jose JB, Tufman A, Drutz HP, Murphy K. Assessment of patient satisfaction with postoperative pain management after ambulatory gynaecologic laparoscopy. J Obstet Gynaecol Can. 2007 Aug;29(8):664-7. doi: 10.1016/s1701-2163(16)32552-x. PMID 17714620
- [Background] Kehlet H, Holte K. Effect of postoperative analgesia on surgical outcome. Br J Anaesth. 2001 Jul;87(1):62-72. doi: 10.1093/bja/87.1.62. No abstract available. PMID 11460814
- [Background] McKay A, Gottschalk A, Ploppa A, Durieux ME, Groves DS. Systemic lidocaine decreased the perioperative opioid analgesic requirements but failed to reduce discharge time after ambulatory surgery. Anesth Analg. 2009 Dec;109(6):1805-8. doi: 10.1213/ANE.0b013e3181be371b. PMID 19923506
- [Background] White PF. The changing role of non-opioid analgesic techniques in the management of postoperative pain. Anesth Analg. 2005 Nov;101(5 Suppl):S5-S22. doi: 10.1213/01.ANE.0000177099.28914.A7. PMID 16334489
- [Background] Koppert W, Weigand M, Neumann F, Sittl R, Schuettler J, Schmelz M, Hering W. Perioperative intravenous lidocaine has preventive effects on postoperative pain and morphine consumption after major abdominal surgery. Anesth Analg. 2004 Apr;98(4):1050-1055. doi: 10.1213/01.ANE.0000104582.71710.EE. PMID 15041597
- [Background] Groudine SB, Fisher HA, Kaufman RP Jr, Patel MK, Wilkins LJ, Mehta SA, Lumb PD. Intravenous lidocaine speeds the return of bowel function, decreases postoperative pain, and shortens hospital stay in patients undergoing radical retropubic prostatectomy. Anesth Analg. 1998 Feb;86(2):235-9. doi: 10.1097/00000539-199802000-00003. PMID 9459225
- [Background] Kaba A, Laurent SR, Detroz BJ, Sessler DI, Durieux ME, Lamy ML, Joris JL. Intravenous lidocaine infusion facilitates acute rehabilitation after laparoscopic colectomy. Anesthesiology. 2007 Jan;106(1):11-8; discussion 5-6. doi: 10.1097/00000542-200701000-00007. PMID 17197840
- [Background] Marret E, Rolin M, Beaussier M, Bonnet F. Meta-analysis of intravenous lidocaine and postoperative recovery after abdominal surgery. Br J Surg. 2008 Nov;95(11):1331-8. doi: 10.1002/bjs.6375. PMID 18844267
- [Background] Gill TM, Feinstein AR. A critical appraisal of the quality of quality-of-life measurements. JAMA. 1994 Aug 24-31;272(8):619-26. PMID 7726894
- [Background] Guyatt GH, Cook DJ. Health status, quality of life, and the individual. JAMA. 1994 Aug 24-31;272(8):630-1. No abstract available. PMID 8057520
- [Background] Watcha MF, Issioui T, Klein KW, White PF. Costs and effectiveness of rofecoxib, celecoxib, and acetaminophen for preventing pain after ambulatory otolaryngologic surgery. Anesth Analg. 2003 Apr;96(4):987-994. doi: 10.1213/01.ANE.0000053255.93270.31. PMID 12651647
- [Background] Myles PS, Hunt JO, Nightingale CE, Fletcher H, Beh T, Tanil D, Nagy A, Rubinstein A, Ponsford JL. Development and psychometric testing of a quality of recovery score after general anesthesia and surgery in adults. Anesth Analg. 1999 Jan;88(1):83-90. doi: 10.1097/00000539-199901000-00016. PMID 9895071
- [Background] Myles PS, Weitkamp B, Jones K, Melick J, Hensen S. Validity and reliability of a postoperative quality of recovery score: the QoR-40. Br J Anaesth. 2000 Jan;84(1):11-5. doi: 10.1093/oxfordjournals.bja.a013366. PMID 10740540
- [Derived] De Oliveira GS Jr, Fitzgerald P, Streicher LF, Marcus RJ, McCarthy RJ. Systemic lidocaine to improve postoperative quality of recovery after ambulatory laparoscopic surgery. Anesth Analg. 2012 Aug;115(2):262-7. doi: 10.1213/ANE.0b013e318257a380. Epub 2012 May 14. PMID 22584558

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited in the preoperative area of the hospital between November 2010 and September 2011.
Pre-assignment Details: All participants were assigned to groups.
Groups:
- Group A (Study Group) Lidocaine: Group A (study group) Lidocaine administration
- Placebo: Group B (control group) will receive the same volume of saline infusion.
Period: Overall Study
Arm/Group | Group A (Study Group) Lidocaine | Placebo
Started | 35 | 35
Completed | 31 | 32
Not Completed | 4 | 3
Not completed — Change to open surgical procedure | 4 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group A (Study Group) Lidocaine | Placebo | Total
Number analyzed (Participants) | 35 | 35 | 70
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 35 | 35 | 70
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.2 (8.6) | 39.1 (9.3) | 38.2 (9.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35 | 35 | 70
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 35 | 35 | 70

OUTCOME MEASURES:

1. Primary Outcome: Quality of Recovery 40 Score
Description: Quality of recovery 40 score on the day after surgery. Scale ranges from a low of 40 (poor recovery) to a high of 200 (good recovery).
Time Frame: 24 hours post surgery
Population: Intent to treat.
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Group A (Study Group) Lidocaine | Placebo
Number analyzed (Participants) | 31 | 32
units on a scale | 175 [160 to 183] | 157.5 [142.5 to 173.5]

2. Secondary Outcome: Opioid Consumption (Morphine Equivalents)
Description: opioid consumption (morphine equivalents)post operatively
Time Frame: 24 hours
Measure: Median (Full Range); unit: mg
Arm/Group | Group A (Study Group) Lidocaine | Placebo
Number analyzed (Participants) | 31 | 32
mg | 20 [0 to 30] | 30 [15 to 35]

ADVERSE EVENTS:
Time Frame: 2 Days
Arm/Group | Group A (Study Group) Lidocaine | Placebo
Serious Adverse Events (participants affected / at risk) | 0/35 | 0/35
Other Adverse Events (participants affected / at risk) | 12/35 | 17/35
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group A (Study Group) Lidocaine (N=35) | Placebo (N=35)
Nausea (Gastrointestinal disorders) | 12 (12) | 17 (17)
Vomiting (Gastrointestinal disorders) | 8 (8) | 10 (10)

LIMITATIONS AND CAVEATS:
Quality of recovery (QOR-40) instrument validation was performed in the in-patient setting and formal validation for the outpatient setting is still lacking.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No